CLINICAL TRIAL: NCT03701815
Title: Assessing the Effect of Multi-disciplinary Lifestyle Medicine Intervention on Brain-derived Neurotrophic Factor Levels Following Stroke
Brief Title: Effect of Lifestyle Changes on BDNF Level After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Collaborators: Stanford University (Other); Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Jeffrey Krauss, Staff Physician, VA Palo Alto Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRU001
Record Dates: First submitted 2018-09-27; First posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Stroke
Keywords: brain-derived neurotrophic factor; exercise; BDNF; lifestyle medicine
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Health; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post-stroke (Experimental): Patients will receive a 12-week lifestyle medicine program.
  Interventions: Behavioral: Wellness in Rehabilitation program

INTERVENTIONS:
Behavioral: Wellness in Rehabilitation program — The 12-week Wellness in Rehabilitation program includes weekly in-person meetings including aerobic exercise, nutrition/cooking training, stress management techniques, education, and group support. A health coach will facilitate continuation of healthy behaviors at home.
  Other Names: Lifestyle Medicine program

SUMMARY:
This is a pilot study to determine whether a lifestyle medicine intervention following stroke may increase levels of Brain-Derived Neurotrophic Factor (BDNF).

DETAILED DESCRIPTION:
This is a substudy of the study entitled "Assessing a Multi-Disciplinary Lifestyle Medicine Intervention Following Stroke," specifically looking at the effects of lifestyle change on brain-derived neurotrophic factor (BDNF). BDNF has emerged as a key facilitator of neuroplasticity to improve motor learning and rehabilitation after stroke. Aerobic exercise has been shown to increase levels of BDNF in multiple parts of the central nervous system and therefore may facilitate neuroplasticity and motor recovery. While BDNF levels appear to be increased for up to 1 hour following a bout of aerobic exercise, it is unclear whether regular aerobic exercise over weeks to months can increase baseline BDNF levels in humans following stroke.

An single nucleotide polymorphism exists on the BDNF gene in 30-50% of the human population that results in an amino acid change from valine (val) to methionine (met) at position 66 (val66met) of the precursor peptide proBDNF. The presence of the met allele results in a 25% reduction in activity-dependent secretion of BDNF in the CNS.

The Wellness in Rehabilitation program at the VA Palo Alto Health Care System is a lifestyle medicine intervention for patients following stroke. It is a 12-week program involving weekly meetings that include exercise (particularly aerobic exercise), nutrition, stress management, education, and group support. Participants are encouraged to perform healthy lifestyle behaviors (i.e. exercise) daily at home, and a health coach calls each patient weekly to support the behavior change process.

Participants in the Wellness in Rehabilitation program who elect to participate in the research study will have blood drawn at baseline, week 6, and week 12. Blood draws will be performed in the morning prior to exercise, and week 6 will additionally include a blood draw within 30 minutes of completing a bout of aerobic exercise. Following completion of the study, plasma BDNF levels (measured as nanograms per milliliter) will then be measured at all 4 time points (baseline, week 6 pre-exercise, week 6 post-exercise, and week 12). In addition, BDNF genotype will be measured using the baseline sample. Participants will also complete bike or treadmill exercise testing at baseline and week 12 to determine pre- and post-program cardiovascular fitness levels (measured as VO2 max and estimated metabolic equivalents), and will also complete a 6-minute walk test. They will be asked to record their exercise daily and will additionally complete the Physical Activity Scale for Individuals with Physical Disabilities at baseline and week 12 time points.

ELIGIBILITY:
Inclusion Criteria:

* History of prior stroke (ischemic or hemorrhagic) or transient ischemic attack
* Ability to ambulate at least 10 feet with minimal to moderate assistance
* Ability to travel to intervention site on a weekly basis.

Exclusion Criteria:

* Cerebral aneurysm
* Concurrent pregnancy
* Serious terminal illnesses (e.g. end stage renal disease, heart failure (class IV), cirrhosis (class C), metastatic cancer)
* Any injury or illness preventing participation in regular aerobic exercise
* Moderate-severe dementia or cognitive decline

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-01-19 (Actual); Primary Completion 2019-01-11 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
BDNF level - Final | Week 12
  Plasma BDNF protein levels, expressed in nanograms per milliliter, measured prior to any exercise upon completion of intervention.

SECONDARY OUTCOMES:
BDNF level - Post-exercise | Week 6
  Plasma BDNF protein levels, expressed in nanograms per milliliter, measured immediately following bout of aerobic exercise.
BDNF Genotype | Baseline
  Genotyping of venous blood samples to determine ValVal, MetMet, and ValMet distribution.
Cardiovascular Fitness - VO2 max | Week 12
  Measured as VO2 max (ml/kg/min).
Cardiovascular Fitness - METs | Week 12
  Measured as estimated metabolic equivalents (kcal/kg/hour).
6-minute Walk Test | Week 12
  Total distance walked 6 minutes on a flat surface.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Krauss, MD, Principal Investigator — VA Palo Alto Health Care System, Stanford University
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided